CLINICAL TRIAL: NCT01048515
Title: The Effect of Caffeine as Endurance Enhancing Drug in the Elderly Following Eight Hour Abstinence From Caffeine Containing Drinks and Foods
Brief Title: The Effect of Caffeine in Elderly Citizen Following Eight Hour Abstinence From Caffeine Containing Drinks & Foods
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herning Hospital (Other)
Responsible Party: Martin Bach Jensen, MD, Ph.d., Surgical Research Department, Herning Hospital, DK-7400 Herning
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MBJ-1
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Healthy; Elderly
Keywords: Caffeine; Physiological Effects of Drugs; Central Nervous System Agents
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caffeine (Experimental)
  Interventions: Drug: Caffeine
- Placebo (Placebo Comparator)
  Interventions: Drug: Caffeine

INTERVENTIONS:
Drug: Caffeine — Caffeine capsule 6 mg/kg given 1 hour before test
  Other Names: Identical looking placebo capsule given 1 hour before test

SUMMARY:
The study investigated the effect of caffeine on physical performance in healthy citizens aged over 70 years following eight hours of abstinence from caffeine containing drinks and foods. The main hypothesis was that 6 mg/kg caffeine would improve cycling endurance at 65% of expected maximal heart rate.

DETAILED DESCRIPTION:
It is well documented that caffeine ingestion increases the endurance of young people exercising at 60%-85% of their maximal oxygen uptake (13;15;47). It also seems to improve endurance as measured by repeated sub-maximal isometric contraction (42), and decreases the rate of perceived exertion during exercise (6;9;46). Typically, doses of approximately 6 mg/kg caffeine were used in these studies.

With a growing number of elderly with a physical active lifestyle and many elderly participating in rehabilitation programs the endurance enhancing effect of caffeine is of increasing interest in this age group. We therefore conducted a study of healthy 75 year old citizens to investigate whether 6 mg/kg caffeine improved physical performance and reduced the perceived effort during work in healthy citizens aged ≥ 70 years. The main hypothesis was that caffeine would improve cycling endurance at 65% of expected maximal heart rate. The study showed that compared to placebo caffeine increased endurance by 25 % (p<0.0001) and isometric sub-maximal strength with 54 % (p<0.0001), reduced perceived exertion after 5 minutes of biking by 11 % (p=0.002), but in 21 of 30 participants there was reduced postural stability (with eyes open). In the above described study participants abstained from caffeine containing drinks and foods for 48 hours prior to each test. Half of the participants reported withdrawal symptoms. Such a long caffeine abstinence period would infer with daily life for many people. We therefore invited the participants from the above study to a repetition of the above study to test whether similar results would be obtained if participants only abstained from caffeine containing drinks and foods for 8 hours prior to each test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy elderly individuals aged over 70 years (Primarily those who previously have participated in an identical study with 48 hour caffeine abstinence)

Exclusion Criteria:

* Dementia or invalidating psychiatric disease
* General debility, angina, or other diseases that would render participation in the test program impossible
* Treatment with beta receptor blocking drugs, calcium-channel blocking drugs, digitalis, or nitroglycerine
* Acute disease and injury
* Diabetes
* Conditions that would contraindicate caffeine ingestion or participation in the test program
* Treatment with medication that interacts with caffeine
* Ingestion of caffeine containing drinks and foods 8 hours before each session

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-02; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Endurance measured on an ergometer bicycle | The tests started 1 h following placebo/caffeine

SECONDARY OUTCOMES:
Isometric endurance (arm flexion) | The tests started 1 h following placebo/caffeine
Isometric maximum arm flexion strength | The tests started 1 h following placebo/caffeine
Fatigue (Borg scale) during ergometer test | After 5 minutes biking and at exhaustion
Postural stability | The tests started 1 h following placebo/caffeine
Reaction time | The tests started 1 h following placebo/caffeine
Walking speed | The tests started 1 h following placebo/caffeine
Biochemistry: lactate, catecholamines, insulin, free fatty acids, glucose | Before intervention; before cycling; after 5 minutes of cycling; and at exhaustion
Withdrawal symptoms | At the end of each test
Side effects | At the end of each test

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Jensen, MD, Ph.d., Principal Investigator — Surgical Research Unit, Department of Surgery P, Aarhus University Hospital
Locations (1):
- Surgical Research Department, Herning, Central Jutland, Denmark

REFERENCES:
- [Background] Norager CB, Jensen MB, Madsen MR, Laurberg S. Caffeine improves endurance in 75-yr-old citizens: a randomized, double-blind, placebo-controlled, crossover study. J Appl Physiol (1985). 2005 Dec;99(6):2302-6. doi: 10.1152/japplphysiol.00309.2005. Epub 2005 Aug 4. PMID 16081625
- [Background] Norager CB, Jensen MB, Weimann A, Madsen MR. Metabolic effects of caffeine ingestion and physical work in 75-year old citizens. A randomized, double-blind, placebo-controlled, cross-over study. Clin Endocrinol (Oxf). 2006 Aug;65(2):223-8. doi: 10.1111/j.1365-2265.2006.02579.x. PMID 16886964